CLINICAL TRIAL: NCT01781858
Title: Study on the Clinical Course Of Pulmonary Embolism
Acronym: SCOPE
Status: Completed | Type: Observational
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Raffaele Pesavento, MD, University of Padova
Other Study IDs: Scope-001
Record Dates: First submitted 2013-01-30; First posted 2013-02-01 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Cardiovascular Diseases; Venous Thromboembolism; Pulmonary Hypertension
Keywords: Pulmonary embolism; Chronic thromboembolic pulmonary hypertension; Venous thromboembolism
MeSH Terms: conditions — Cardiovascular Diseases; Venous Thromboembolism; Hypertension, Pulmonary; Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- pulmonary embolism: Consecutive outpatients and inpatients with first episode of acute pulmonary embolism

SUMMARY:
The course of both pulmonary embolism (PE) and one of its more relevant late complications, i.e. chronic thromboembolic pulmonary hypertension (CTEPH) is still substantially unknown.

Recent evidence has shown that the incidence of CTEPH is higher than previously believed, but this has not been confirmed by other studies. A clear link between PE and CTEPH has been questioned by some experts. A great number of patients affected by PE persistently have residual chronic thromboembolic material the meaning of which is a matter of debate. The evidence sustaining a link between chronic residual PE and subsequent PE recurrences or CTEPH is insufficient.

Thus, a nationwide, multicentre, prospective cohort study was designed with the following aims:

1. to ascertain the incidence of symptomatic CTEPH after a first episode of acute PE;
2. to ascertain the incidence of venous thromboembolic (VTE) recurrences after a first episode of acute PE;
3. to evaluate whether a relation exists between chronic residual PE and CTEPH
4. to evaluate whether a relation exists between chronic residual PE and VTE recurrences;
5. to evaluate whether a relation exists between persistent right ventricular dysfunction and CTEPH;
6. to evaluate whether a relation exists between persistent right ventricular dysfunction and PE recurrences.

For each enrolling centre, consecutive outpatients or inpatients with an objectively diagnosed first acute PE episode are considered eligible.

DETAILED DESCRIPTION:
All patients enrolled in the study received a diagnosis of PE by means of chest CT scan, lung scanning or pulmonary angiography. All patients should undergo an echocardiographic examination during the acute phase of PE, when this is possible. All patients will be treated according to current international guidelines and local protocols. All surviving patients will receive an echocardiographic examination after 6 weeks and 6 months. All surviving patients will receive a perfusional pulmonary scintigraphy at 6 months and be subsequently followed up every 6 months for at least 3 years.

In case of clinical suspicion of VTE recurrence a diagnostic procedure will be performed in order to confirm the recurrent VTE episode ( Chest CT scan, lung scan, Pulmonary angiography, compressive ultrasound, phlebography, vein CT scan).

In case of clinical suspicion of CTEPH, a further diagnostic workup will be performed, consisting in echocardiography, ventilation/perfusion lung scanning, multidetector chest CT scanning, and pulmonary angiography, with direct measurement of the pulmonary-artery pressure.

The extension of pulmonary embolism during the acute phase will be graded according to a standardized scoring system by local investigators while the extension of chronic residual pulmonary embolism will be graded according to a standardized scoring system ( Meyer score) by both local investigators and an independent committee. All outcome events will be centrally adjudicated by an independent committee.

All clinical data ( initial data on medical history, clinical symptoms, presence of risk factors, diagnoses, diagnostic tests results, treatment type and duration, outcome events and other) will be collected by the local investigators in an electronic medical database. Related data will be sent to the coordinating centre on a regular basis. All recruiting centres will be regularly monitored by the coordinating Centre.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive Outpatients/Inpatients with acute first episode of acute pulmonary embolism

Exclusion Criteria:

* Pregnancy
* Age < 18 years
* expected survival < 2 years
* previous episodes of VTE
* need for anticoagulation for reasons other than VTE
* preexisting severe cardiac or pulmonary diseases
* preexisting diseases that could cause non thromboembolic pulmonary hypertension
* Patients geographically inaccessible for follow up
* Low compliance to anticoagulant therapy and planned diagnostic work-up
* Refusal to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive outpatients or inpatients with an objective diagnosis of first acute PE episode.
Sampling Method: Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2008-01; Primary Completion 2014-05 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Incidence of chronic thromboembolic pulmonary hypertension | within 3 years

SECONDARY OUTCOMES:
Incidence of recurrent venous thromboembolic events | within 3 years

OTHER OUTCOMES:
Incidence of all-cause mortality | within 3 years
Incidence of Pulmonary Embolism - related mortality | within 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele Pesavento, MD, Study Director — University of Padova; Paolo Prandoni, MD,PHD, Study Chair — University of Padova; Antonio Pagnan, MD, Study Chair — University of Padova; Gualtiero Palareti, MD, Study Chair — University of Bologna; Antonio Palla, MD, Study Chair — University of Pisa; Vittorio Pengo, MD, Study Chair — University of Padova; Franco Piovella, MD, Study Chair — University of Pavia - Italy

REFERENCES:
- [Background] Pengo V, Lensing AW, Prins MH, Marchiori A, Davidson BL, Tiozzo F, Albanese P, Biasiolo A, Pegoraro C, Iliceto S, Prandoni P; Thromboembolic Pulmonary Hypertension Study Group. Incidence of chronic thromboembolic pulmonary hypertension after pulmonary embolism. N Engl J Med. 2004 May 27;350(22):2257-64. doi: 10.1056/NEJMoa032274. PMID 15163775
- [Background] Becattini C, Agnelli G, Pesavento R, Silingardi M, Poggio R, Taliani MR, Ageno W. Incidence of chronic thromboembolic pulmonary hypertension after a first episode of pulmonary embolism. Chest. 2006 Jul;130(1):172-5. doi: 10.1378/chest.130.1.172. PMID 16840398
- [Background] Lang IM, Pesavento R, Bonderman D, Yuan JX. Risk factors and basic mechanisms of chronic thromboembolic pulmonary hypertension: a current understanding. Eur Respir J. 2013 Feb;41(2):462-8. doi: 10.1183/09031936.00049312. Epub 2012 Jun 14. PMID 22700839
- [Background] Prandoni P, Noventa F, Ghirarduzzi A, Pengo V, Bernardi E, Pesavento R, Iotti M, Tormene D, Simioni P, Pagnan A. The risk of recurrent venous thromboembolism after discontinuing anticoagulation in patients with acute proximal deep vein thrombosis or pulmonary embolism. A prospective cohort study in 1,626 patients. Haematologica. 2007 Feb;92(2):199-205. doi: 10.3324/haematol.10516. PMID 17296569
- [Background] Verso M, Agnelli G, Ageno W, Imberti D, Moia M, Palareti G, Pistelli R, Cantone V; MASTER investigators. Long-term death and recurrence in patients with acute venous thromboembolism: the MASTER registry. Thromb Res. 2012 Sep;130(3):369-73. doi: 10.1016/j.thromres.2012.04.003. Epub 2012 May 13. PMID 22583838
- [Background] Cosmi B, Nijkeuter M, Valentino M, Huisman MV, Barozzi L, Palareti G. Residual emboli on lung perfusion scan or multidetector computed tomography after a first episode of acute pulmonary embolism. Intern Emerg Med. 2011 Dec;6(6):521-8. doi: 10.1007/s11739-011-0577-8. Epub 2011 Apr 3. PMID 21461909
- [Background] Alhadad A, Miniati M, Alhadad H, Gottsater A, Bajc M. The value of tomographic ventilation/perfusion scintigraphy (V/PSPECT) for follow-up and prediction of recurrence in pulmonary embolism. Thromb Res. 2012 Dec;130(6):877-81. doi: 10.1016/j.thromres.2012.09.002. Epub 2012 Sep 29. PMID 23026380
- [Background] Poli D, Miniati M. The incidence of recurrent venous thromboembolism and chronic thromboembolic pulmonary hypertension following a first episode of pulmonary embolism. Curr Opin Pulm Med. 2011 Sep;17(5):392-7. doi: 10.1097/MCP.0b013e328349289a. PMID 21743331
- [Background] Poli D, Grifoni E, Antonucci E, Arcangeli C, Prisco D, Abbate R, Miniati M. Incidence of recurrent venous thromboembolism and of chronic thromboembolic pulmonary hypertension in patients after a first episode of pulmonary embolism. J Thromb Thrombolysis. 2010 Oct;30(3):294-9. doi: 10.1007/s11239-010-0452-x. PMID 20157841
- [Background] Miniati M, Monti S, Bottai M, Scoscia E, Bauleo C, Tonelli L, Dainelli A, Giuntini C. Survival and restoration of pulmonary perfusion in a long-term follow-up of patients after acute pulmonary embolism. Medicine (Baltimore). 2006 Sep;85(5):253-262. doi: 10.1097/01.md.0000236952.87590.c8. PMID 16974210
- [Background] Nijkeuter M, Sohne M, Tick LW, Kamphuisen PW, Kramer MH, Laterveer L, van Houten AA, Kruip MJ, Leebeek FW, Buller HR, Huisman MV; Christopher Study Investigators. The natural course of hemodynamically stable pulmonary embolism: Clinical outcome and risk factors in a large prospective cohort study. Chest. 2007 Feb;131(2):517-23. doi: 10.1378/chest.05-2799. PMID 17296656
- [Background] Nijkeuter M, Hovens MM, Davidson BL, Huisman MV. Resolution of thromboemboli in patients with acute pulmonary embolism: a systematic review. Chest. 2006 Jan;129(1):192-7. doi: 10.1378/chest.129.1.192. PMID 16424432
- [Background] Pepke-Zaba J, Delcroix M, Lang I, Mayer E, Jansa P, Ambroz D, Treacy C, D'Armini AM, Morsolini M, Snijder R, Bresser P, Torbicki A, Kristensen B, Lewczuk J, Simkova I, Barbera JA, de Perrot M, Hoeper MM, Gaine S, Speich R, Gomez-Sanchez MA, Kovacs G, Hamid AM, Jais X, Simonneau G. Chronic thromboembolic pulmonary hypertension (CTEPH): results from an international prospective registry. Circulation. 2011 Nov 1;124(18):1973-81. doi: 10.1161/CIRCULATIONAHA.110.015008. Epub 2011 Oct 3. PMID 21969018
- [Background] Korkmaz A, Ozlu T, Ozsu S, Kazaz Z, Bulbul Y. Long-term outcomes in acute pulmonary thromboembolism: the incidence of chronic thromboembolic pulmonary hypertension and associated risk factors. Clin Appl Thromb Hemost. 2012 Jun;18(3):281-8. doi: 10.1177/1076029611431956. Epub 2012 Jan 23. PMID 22275389
- [Background] Wilkens H, Lang I, Behr J, Berghaus T, Grohe C, Guth S, Hoeper MM, Kramm T, Kruger U, Langer F, Rosenkranz S, Schafers HJ, Schmidt M, Seyfarth HJ, Wahlers T, Worth H, Mayer E. Chronic thromboembolic pulmonary hypertension (CTEPH): updated Recommendations of the Cologne Consensus Conference 2011. Int J Cardiol. 2011 Dec;154 Suppl 1:S54-60. doi: 10.1016/S0167-5273(11)70493-4. PMID 22221974
- [Background] Willemink MJ, van Es HW, Koobs L, Morshuis WJ, Snijder RJ, van Heesewijk JP. CT evaluation of chronic thromboembolic pulmonary hypertension. Clin Radiol. 2012 Mar;67(3):277-85. doi: 10.1016/j.crad.2011.09.012. Epub 2011 Nov 25. PMID 22119298
- [Background] Ley S, Ley-Zaporozhan J, Pitton MB, Schneider J, Wirth GM, Mayer E, Duber C, Kreitner KF. Diagnostic performance of state-of-the-art imaging techniques for morphological assessment of vascular abnormalities in patients with chronic thromboembolic pulmonary hypertension (CTEPH). Eur Radiol. 2012 Mar;22(3):607-16. doi: 10.1007/s00330-011-2290-4. Epub 2011 Sep 27. PMID 21947513
- [Background] Piazza G, Goldhaber SZ. Chronic thromboembolic pulmonary hypertension. N Engl J Med. 2011 Jan 27;364(4):351-60. doi: 10.1056/NEJMra0910203. No abstract available. PMID 21268727
- [Background] Marti D, Gomez V, Escobar C, Wagner C, Zamarro C, Sanchez D, Sam A, Briongos S, Gaudo J, Sueiro A, Jimenez D. [Incidence of symptomatic and asymptomatic chronic thromboembolic pulmonary hypertension]. Arch Bronconeumol. 2010 Dec;46(12):628-33. doi: 10.1016/j.arbres.2010.07.012. Spanish. PMID 20926172
- [Background] Surie S, Gibson NS, Gerdes VE, Bouma BJ, van Eck-Smit BL, Buller HR, Bresser P. Active search for chronic thromboembolic pulmonary hypertension does not appear indicated after acute pulmonary embolism. Thromb Res. 2010 May;125(5):e202-5. doi: 10.1016/j.thromres.2009.12.016. Epub 2010 Jan 20. PMID 20085846
- [Background] Klok FA, van Kralingen KW, van Dijk AP, Heyning FH, Vliegen HW, Huisman MV. Prospective cardiopulmonary screening program to detect chronic thromboembolic pulmonary hypertension in patients after acute pulmonary embolism. Haematologica. 2010 Jun;95(6):970-5. doi: 10.3324/haematol.2009.018960. Epub 2010 Jan 6. PMID 20053871
- [Derived] Pesavento R, Filippi L, Palla A, Visona A, Bova C, Marzolo M, Porro F, Villalta S, Ciammaichella M, Bucherini E, Nante G, Battistelli S, Muiesan ML, Beltramello G, Prisco D, Casazza F, Ageno W, Palareti G, Quintavalla R, Monti S, Mumoli N, Zanatta N, Cappelli R, Cattaneo M, Moretti V, Cora F, Bazzan M, Ghirarduzzi A, Frigo AC, Miniati M, Prandoni P; SCOPE Investigators. Impact of residual pulmonary obstruction on the long-term outcome of patients with pulmonary embolism. Eur Respir J. 2017 May 25;49(5):1601980. doi: 10.1183/13993003.01980-2016. Print 2017 May. PMID 28546279